CLINICAL TRIAL: NCT00111670
Title: A Randomized, Double-blind Study of the Effect of the DPP-IV Inhibitor on HbA1c and Safety in Patients With Type 2 Diabetes
Brief Title: A Study of DPP-IV Inhibitor in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM18102
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: DPP-IV Inhibitor
- 2 (Experimental)
  Interventions: Drug: DPP-IV Inhibitor
- 3 (Experimental)
  Interventions: Drug: DPP-IV Inhibitor
- 4 (Experimental)
  Interventions: Drug: DPP-IV Inhibitor
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DPP-IV Inhibitor — Escalating doses po bid or qd
  Arms: 1; 2; 3; 4
Drug: Placebo — po bid or qd
  Arms: 5

SUMMARY:
This study will assess the efficacy, safety and tolerability of DPP-IV Inhibitor compared to placebo in patients with type 2 diabetes. The anticipated time on study treatment is < 3 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-75 years of age;
* type 2 diabetes diagnosed >=1 month before screening;
* no previous treatment, or previous treatment with no more than 2 oral medications.

Exclusion Criteria:

* type 1 diabetes;
* type 2 diabetes treated with insulin or a PPAR gamma agonist during the 3 months before screening;
* patients who are pregnant, breastfeeding or not using a reliable contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2005-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbAlc\n\n | Week 12

SECONDARY OUTCOMES:
Absolute change in FPG and absolute/relative change in insulin sensitivity, beta-cell-function, lipid profile, response rate | Week 12
AEs, vital signs, laboratory tests, body weight, waist/hip ratio, ECG\n | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- United States (18):
  - Salinas, California
  - Clearwater, Florida
  - Hialeah, Florida
  - Pembroke Pines, Florida
  - Blue Ridge, Georgia
  - Aurora, Illinois
  - Elkton, Maryland
  - Oxon Hill, Maryland
  - Troy, Michigan
  - Pahrump, Nevada
  - Cincinnati, Ohio
  - Portland, Oregon
  - Warminster, Pennsylvania
  - Dallas, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Virginia Beach, Virginia
- Bulgaria (2):
  - Rousse
  - Sofia
- San José, Costa Rica
- Tartu, Estonia
- Latvia (2):
  - Ogre
  - Riga
- Lithuania (2):
  - Klaipėda
  - Vilnius
- Mexico (5):
  - Chihuahua City
  - Guadalajara
  - Mexico City
  - Monterrey
  - Pachuca
- Ponce, Puerto Rico
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Ploieşti
  - Târgu Mureş